CLINICAL TRIAL: NCT01757769
Title: Effectiveness and Safety of Silodosin in the Treatment of LUTS in Patients With Benign Prostatic Hyperplasia: a European Phase IV Clinical Study. The Silodosin in Real-life Evaluation Study
Brief Title: Effectiveness and Safety of Silodosin in the Treatment of Benign Prostatic Hyperplasia
Acronym: SiRE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: RECORDATI GROUP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMD 3213 IT-CL 0376; 2011-000045-20 (EudraCT Number)
Record Dates: First submitted 2012-12-21; First posted 2012-12-31 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Lower urinary tract symptoms; benign prostatic hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — silodosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Silodosin (Experimental): Silodosin capsule 8 mg daily for 24 weeks
  Interventions: Drug: Silodosin

INTERVENTIONS:
Drug: Silodosin — 8 mg daily for 24 weeks

SUMMARY:
The purpose of this study is to confirm in a larger population in Europe the effectiveness and safety observed with silodosin in previous clinical trials.

DETAILED DESCRIPTION:
The objective of the study is to confirm in a larger and less selected population ("real life conditions") the positive risk-benefit balance observed with silodosin in double-blind, randomised clinical trials.

The following aspects will be evaluated:

* the effects on lower urinary tract symptoms (LUTS), by means of the International Prostate Symptoms Score (IPSS) questionnaire
* the effect on the most frequent and bothersome symptoms, by means of International Continence Society (ICS)-male questionnaire
* the effects on Quality of Life (QoL) due to urinary symptoms
* the safety profile
* the adherence to therapy
* the patient satisfaction with treatment The effectiveness and safety of the drug will be investigated also in different subgroups of subjects according to age, severity of the disease, concomitant disease and medications.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Benign Prostatic Hyperplasia (BPH) by the urologist;
* Male subjects aged 60 years or older;
* IPSS total score equal or more than 12 at Visit 1 (Screening) and 2 (Baseline);
* Able to comply with protocol procedures;
* Written informed consent obtained before beginning any investigational procedures.

Exclusion Criteria:

* Hypersensitivity to the active substance or to any of the excipients;
* Patients for whom cataract surgery is scheduled;
* History of orthostatic hypotension or syncope;
* Moderate or severe renal impairment (CLCR <50 ml/min, as estimated by the Cockcroft Gault formula);
* Severe hepatic impairment;
* Concomitant use of other α-adrenoreceptor antagonists or natural/herbal products known to have an effect on LUTS (e.g. saw palmetto - serenoa serrulate/repens) . Patients already on treatment with those drugs may be enrolled after a 4 week wash-out period before Visit 2 (baseline);
* Concomitant use with potent cytochrome P450 3A4 inhibitors, such as ketoconazole, itraconazole or ritonavir (possible pharmacokinetic interaction);
* Prostate cancer;
* History of prostate or bladder neck surgery, including transurethral prostatectomy, TUNA, laser or other minimally invasive therapy;
* Active urinary tract infection;
* Acute or recurrent prostatitis (more than 3 times in the last year);
* History of neurological disease that may affect bladder function;
* Unstable cardiovascular or cerebrovascular disease (including acute myocardial infarction, unstable angina pectoris, by-pass, percutaneous transluminal coronary angioplasty, congestive heart failure class III-IV, stroke, transient ischemic attack and episodes of cardiac arrhythmia requiring treatment in the last 6 months);
* History or current evidence of drug or alcohol abuse within the last 12 months;
* Participation in a study involving the administration of an investigational compound within the past 30 days;
* Any other condition which, in the investigator's judgement, renders the subject unable to complete the study or increases the risk to the subject or which prevents optimal participation in achieving the objectives of the study.

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1036 (Actual)
Dates: Start 2011-05; Primary Completion 2013-03 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to evaluate the effects of silodosin on LUTS in terms of IPSS response rate (decrease from baseline ≥ 25% in the IPSS total score) | 6 months o treatment

SECONDARY OUTCOMES:
Change from baseline in IPSS total score | 4, 12, 24 weeks of treatment

OTHER OUTCOMES:
Percentage of subjects improving each symptom of the ICS (International Continence Society) male questionnaire as compared to baseline; to evaluate the effect of silodosin on the most frequent and bothersome symptoms | 6 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R Chapple, MD, Study Chair — Urology Department, Royal Hallamshire Hospital, University of Sheffield, Glossop Road, Sheffield, S10 2JF, UK
Locations (1):
- Vita e Salute University, Department of Urology, Istituto Scientifico Ospedale San Raffaele, Milan, Italy

REFERENCES:
- [Background] Armitage P., Berry G., Matthews JNS Statistical Methods In Medical Research, 4th Ed. Wiley Blackwell Science 2001
- [Background] Barkin J, Roehrborn CG, Siami P, Haillot O, Morrill B, Black L, Montorsi F; CombAT Study Group. Effect of dutasteride, tamsulosin and the combination on patient-reported quality of life and treatment satisfaction in men with moderate-to-severe benign prostatic hyperplasia: 2-year data from the CombAT trial. BJU Int. 2009 Apr;103(7):919-26. doi: 10.1111/j.1464-410X.2009.08196.x. Epub 2009 Feb 23. PMID 19239460
- [Background] Barry MJ, Fowler FJ Jr, O'Leary MP, Bruskewitz RC, Holtgrewe HL, Mebust WK, Cockett AT. The American Urological Association symptom index for benign prostatic hyperplasia. The Measurement Committee of the American Urological Association. J Urol. 1992 Nov;148(5):1549-57; discussion 1564. doi: 10.1016/s0022-5347(17)36966-5. PMID 1279218
- [Background] Barry MJ, Williford WO, Chang Y, Machi M, Jones KM, Walker-Corkery E, Lepor H. Benign prostatic hyperplasia specific health status measures in clinical research: how much change in the American Urological Association symptom index and the benign prostatic hyperplasia impact index is perceptible to patients? J Urol. 1995 Nov;154(5):1770-4. doi: 10.1016/s0022-5347(01)66780-6. PMID 7563343
- [Background] Black L, Grove A, Morrill B. The psychometric validation of a US English satisfaction measure for patients with benign prostatic hyperplasia and lower urinary tract symptoms. Health Qual Life Outcomes. 2009 Jun 19;7:55. doi: 10.1186/1477-7525-7-55. PMID 19545384
- [Background] Chapple CR, Montorsi F, Tammela TL, Wirth M, Koldewijn E, Fernandez Fernandez E; European Silodosin Study Group. Silodosin therapy for lower urinary tract symptoms in men with suspected benign prostatic hyperplasia: results of an international, randomized, double-blind, placebo- and active-controlled clinical trial performed in Europe. Eur Urol. 2011 Mar;59(3):342-52. doi: 10.1016/j.eururo.2010.10.046. Epub 2010 Nov 10. PMID 21109344
- [Background] de la Rosette J, Alivizatos G, Madersbacher S, Rioja Sanz C, Nordling J, Emberton M, Gravas S, Michel MC, Oelke M. Guidelines on benign prostatic hyperplasia. European Association Urolology 2009
- [Background] Donovan JL, Abrams P, Peters TJ, Kay HE, Reynard J, Chapple C, De La Rosette JJ, Kondo A. The ICS-'BPH' Study: the psychometric validity and reliability of the ICSmale questionnaire. Br J Urol. 1996 Apr;77(4):554-62. doi: 10.1046/j.1464-410x.1996.93013.x. PMID 8777617
- [Background] Donovan JL, Brookes ST, de la Rosette JJ, Peters TJ, Porru D, Kondo A, Dabhoiwala N, Millard R, Bosch R, Nordling J, Matos Ferreira A, Hofner K, Mostafid H, Walter S, Nissenkorn I, Frimodt Moller C, Mendes Silva M, Chapple C, Abrams P. The responsiveness of the ICSmale questionnaire to outcome: evidence from the ICS-'BPH' study. BJU Int. 1999 Feb;83(3):243-8. doi: 10.1046/j.1464-410x.1999.00930.x. PMID 10233487
- [Background] Gisolf KW, van Venrooij GE, Eckhardt MD, Boon TA. Analysis and reliability of data from 24-hour frequency-volume charts in men with lower urinary tract symptoms due to benign prostatic hyperplasia. Eur Urol. 2000 Jul;38(1):45-52. doi: 10.1159/000020251. PMID 10859441
- [Background] Marks LS, Gittelman MC, Hill LA, Volinn W, Hoel G. Rapid efficacy of the highly selective alpha1A-adrenoceptor antagonist silodosin in men with signs and symptoms of benign prostatic hyperplasia: pooled results of 2 phase 3 studies. J Urol. 2009 Jun;181(6):2634-40. doi: 10.1016/j.juro.2009.02.034. Epub 2009 Apr 16. PMID 19371887
- [Background] Michel M. The Pharmacological profile of the a1A-Adrenoceptor antagonist silodosin. Eur Urol Suppl. 9 (2010) 486 - 490
- [Background] Oelke M, Bachmann A, Descazeaud A, Emberton M, Gravas S, Michel MC, N'dow J, Nordling J, de la Rosette JJ; European Association of Urology. EAU guidelines on the treatment and follow-up of non-neurogenic male lower urinary tract symptoms including benign prostatic obstruction. Eur Urol. 2013 Jul;64(1):118-40. doi: 10.1016/j.eururo.2013.03.004. Epub 2013 Mar 13. PMID 23541338
- [Background] Peters TJ, Donovan JL, Kay HE, Abrams P, de la Rosette JJ, Porru D, Thuroff JW. The International Continence Society "Benign Prostatic Hyperplasia" Study: the botherosomeness of urinary symptoms. J Urol. 1997 Mar;157(3):885-9. PMID 9072592